CLINICAL TRIAL: NCT05045274
Title: The Effect of Early Administration of Dapagliflozin in ST Elevation Myocardial Infarction Patients Presenting With Left Ventricular Systolic Dysfunction
Brief Title: The Effect of Early Administration of Dapagliflozin in STEMI Patients With LV Systolic Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, George William Agban, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAgban
Record Dates: First submitted 2021-08-26; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Dysfunction, Left | interventions — dapagliflozin; Aspirin; Ticagrelor; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Adrenergic beta-Antagonists; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dapagliflozin (Active Comparator): (a) Dapagliflozin 10 mg once daily within 24 hours after PPCI for 3 month
  Interventions: Drug: Dapagliflozin 10Mg Tab
- conventional therapy (Placebo Comparator): 1. Reperfusion therapy: primary percutaneous coronary intervention (PPCI) after DAPT loading (aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally) in the ambulance or emergency department upon diagnosis.
  2. Anti-ischemic treatment: DAPT, SC-anticoagulation, beta blockers, statin or others will be individualized according to the patient condition.
  3. Anti-failure treatment: Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — 1. Dapagliflozin: It will be given in a dose of 10 mg once daily within 24 hours after PPCI.
  2. Reperfusion therapy: primary percutaneous coronary intervention (PPCI) after DAPT loading (aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally) in the ambulance or emergency department upon diagnosis.
  3. Anti-ischemic treatment: DAPT, SC-anticoagulation, beta blockers, statin or others will be individualized according to the patient condition.
  4. Anti-failure treatment: Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
  Other Names: aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally; DAPT, SC-anticoagulation, beta blockers, statin; Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
  Arms: dapagliflozin
Drug: Placebo — 1. Reperfusion therapy: primary percutaneous coronary intervention (PPCI) after DAPT loading (aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally) in the ambulance or emergency department upon diagnosis.
  2. Anti-ischemic treatment: DAPT, SC-anticoagulation, beta blockers, statin or others will be individualized according to the patient condition.
  3. Anti-failure treatment: Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
  Other Names: aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally; DAPT, SC-anticoagulation, beta blockers, statin; Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
  Arms: conventional therapy

SUMMARY:
300 STIMI patients with LV systolic dysfunction will be divided into two equal groups (Group I (Study arm, n=150); will receive dapagliflozin plus conventional therapy and group (II) Control arm (n=150); will receive conventional therapy only to detect an improvement in the LVEF by ≥ 5

DETAILED DESCRIPTION:
300 STIMI patients with LV systolic dysfunction will be randomly divided into two equal groups (Group I (Study arm, n=150); will receive

1. Reperfusion therapy: primary percutaneous coronary intervention (PPCI) after DAPT loading (aspirin 300 mg and either clopidogrel 600mg or ticagrelor 180 mg orally) in the ambulance or emergency department upon diagnosis.
2. Anti-ischemic treatment: DAPT, SC-anticoagulation, beta blockers, statin or others will be individualized according to the patient condition.
3. Anti-failure treatment: Angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, mineralocorticoid receptor antagonists, other diuretics will be added in case of volume overload.
4. Dapagliflozin: It will be given in a dose of 10 mg once daily within 24 hours after PPCI.

Group (II) Control arm (n=150); will receive

1. Reperfusion therapy: as in study arm
2. Anti-ischemic treatment: as in study arm.
3. Anti-failure treatment: as in study arm. LV echocardiographic analysis for both groups at baseline and 3 month follow up by 2D Echocardiography to assess: LVEF by simpson method Diastolic function LV diameter and volume. LA volume index. LV mass index. Severity of MR.

Laboratory investigation substudy analysis:

50 patients from either group will undergo NT-proBNP at baseline and after 3 month follow up.

Clinical outcomes:

Patients will be followed up in a deducted outpatient clinic for assessment of clinical outcomes either by phone cell or clinic visits at 3 month.

Patients will be assessed for the following clinical parameters:

I. Composite of CV death and rehospitalization of HF. II. Individual component at composite end points. III. Reinfarction or readmission for ACS and target lesion revascularization.

Research outcome measures:

a. Primary (main):

1. The improvement in the LVEF (≥ 5%) using biplane simpson method echocardiography.

a. Secondary (subsidiary):

1. Echocardiographic parameters at 3 month follow up.

   1. Changes in LV remodeling.
   2. Changes in diastolic function
   3. Changes in LA volume index.
   4. Changes in LV mass index.
2. Laboratory investigations. Changes of the NT-proBNP from baseline to 3 month follow up
3. Clinical outcomes at 3month. I. Composite of CV death and rehospitalization of HF. II. Individual component at composite end points. III. Reinfarction or readmission for ACS and target lesion revascularization.

ELIGIBILITY:
Inclusion Criteria:

* 1st time STEMI within 24 hours undergoing PPCI. (Chest pain > 30 minutes and ST segment elevation in more than one lead, include the definition of MI with a reference: Third universal definition of MI. (published at ESC Clinical Practice Guidelines 2012).
* LVEF less than 50%.
* eGFR ≥20 mL/min/1.73 m2.

Exclusion Criteria:

* Patients less than 18 years old.
* T1D (Type I diabetes mellitus).
* Hemodynamically unstable.
* Cardiogenic shock (clinical syndrome of tissue hypoperfusion resulting from cardiac dysfunction).
* History of chronic symptomatic HF with a prior hHF within last year
* Patients on dialysis.
* Serious hypersensitivity to dapagliflozin (eg, anaphylaxis, angioedema).
* Pregnant or lactating women.
* Sever hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic parameter | 3 month follow up
  The improvement in the LVEF (≥ 5%) using biplane simpson method echocardiography

SECONDARY OUTCOMES:
Changes in LV remodeling | 3 month follow up
  using echocardiography
Changes in diastolic function | 3 month follow up
  using mitral Inflow Patterns electrocardiography
Changes in LA volume index | 3 month follow up
  using by the biplane area-length method from apical 4- and 2-chamber views electrocardiography
Changes in LV mass index. | 3 month follow up
  using by linear method electrocardiography
Laboratory investigations. | 3 month follow up
  Changes of the NT-proBNP from baseline to 3 month follow up
CV death and rehospitalization of HF | 3 month follow up
  Composite of CV death and rehospitalization of HF
Individual component at composite end points. | 3 month follow up
  Composite of CV death or rehospitalization of HF
ACS | 3 month follow up
  Reinfarction or readmission for ACS and target lesion revascularization.